CLINICAL TRIAL: NCT01175694
Title: Phase II Study - Dose Optimization PDR/HDR Brachytherapy Alone for Early Breast Cancer
Brief Title: Dose Optimization for Pulsed-dose-rate (PDR)/High-dose-rate (HDR) Brachytherapy Alone for Early Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Vratislav Strnad, MD, Prof., University Hospital Erlangen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brachy-APBI-03
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
Keywords: Brachytherapy; APBI; dose modification; local recurrences; side effects; cosmetic result
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brachytherapy (Active Comparator): Interstitial multicatheter brachytherapy
  Interventions: Radiation: Interstitial multicatheter brachytherapy

INTERVENTIONS:
Radiation: Interstitial multicatheter brachytherapy — Interstitial PDR- and HDR-brachytherapy up to 50 Gy-eq
  Other Names: APBI

SUMMARY:
Accelerated partial breast irradiation (APBI) leads to a equivalent local control rate with lower toxicity as external beam irradiation (EBI) after breast conserving surgery (BCS) in a highly selected subgroup of patients with low risk invasive carcinoma and low risk duct carcinoma in-situ (DCIS). The goal of this trial is to assess the role of a modified dose of pulsed-dose-rate (PDR) and high-dose-rate (HDR) brachytherapy alone as Accelerated Partial Breast Irradiation (APBI) in a defined low-risk group of invasive breast cancer or ductal carcinoma in situ concerning local failure (all ipsilateral local recurrences), in particular regarding the local recurrences, the toxicity and for the cosmetic result. It is a phase II study. According to study protocol altogether 200 female patients will be treated.

DETAILED DESCRIPTION:
Focus of this trial is to assess the role a modified dose of PDR- and HDR-brachytherapy as Accelerated Partial Breast Irradiation (APBI) alone in a defined low-risk group of invasive breast cancer or ductal carcinoma in situ concerning local failure(all ipsilateral local recurrences, in particular regarding the local recurrences, the toxicity and for the cosmetic result.

ELIGIBILITY:
Inclusion criteria

* Stage 0, I or II breast cancer.
* Invasive ductal, papillary, mucinous, tubular, medullary or lobular carcinoma.
* Ductal carcinoma in situ (DCIS) alone.
* No lymph invasion (L0) and no hemangiosis (V0).
* Lesions of < 3 cm diameter, histopathologically assured.
* pN0 (a minimum of 6 nodes in specimen, or a negative sentinel node is acceptable).
* M0.
* Clear resection margins at least 2 mm in any direction; by lobular histology or DCIS histology only the resection margins must be clear at least 5 mm.
* For DCIS only: lesions must be classified as low or intermediate risk group
* Unifocal and unicentric DCIS or breast cancer.
* Age > 50 years.
* Time interval from final definitive breast surgical procedure to the start of external beam therapy or to brachytherapy is less than 12 weeks (84 days). If patients receive chemotherapy the radiotherapy can be started before systemic treatment (within 12 weeks). The radiation therapy can be also given in the interval between the chemotherapy courses. It is also possible to start radiation therapy after chemotherapy is completed according local protocols as soon as possible within 4 weeks after chemotherapy.
* Signed study-specific consent form

Exclusion Criteria:

* Stage III or IV breast cancer.
* Surgical margins that cannot be microscopically assessed.
* Extensive intraductal component (EIC).
* Paget's disease or pathological skin involvement.
* Synchronous or previous breast cancer.
* Prior malignancy (< 5 years prior to enrollment in study) except non-melanoma skin cancer or cervical carcinoma International Federation of Gynecology and Obstetrics (FIGO) 0 and I if patient is continuously disease-free.
* Pregnant or lactating women.
* Collagen vascular disease.
* The presence of congenital diseases with increased radiation sensitivity, for example Ataxia telangiectatic or similar.
* Psychiatric disorders.
* Patient with breast deemed technically unsatisfactory for brachytherapy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
local control rates | five years

SECONDARY OUTCOMES:
late side effects | 5 years
  to assess the incidence and severity of acute and late side effects of brachytherapy

CONTACTS AND LOCATIONS:
Overall Officials: Vratislav Strnad, MD, Prof., Principal Investigator — University Hospital Erlangen
Locations (1):
- Dept. of Radiation Oncology, University Hospital Erlangen, Erlangen, Germany